CLINICAL TRIAL: NCT06918262
Title: An Observational Clinical Study to Evaluate the Role of MRD in the Prediction of Local Therapy in Patients With Oligometastatic Breast Cancer.
Brief Title: Observational Clinical Study on Role of MRD in Predicting Local Therapy in Oligometastatic Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 24K013-001
Record Dates: First submitted 2025-03-31; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; MRD
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: local treatment — Tumour somatic mutations were identified by 1021 panel sequencing of tumour tissues from cancer patients, and up to 20 mutations were selected as follow-up monitoring loci based on the tumour somatic variants of the patients, and a personalised panel was designed and customised.Post-operative blood from patients was analysed for recurrence risk stratification and drug indications using a combination of personalised panel and a cancer-specific core panel (~5 kb) stacked on top of each other. The postoperative blood of patients was subjected to cfDNA targeted capture and ultra-high depth NGS sequencing (>100,000×) to analyse the status of the surveillance loci in the peripheral blood for recurrence risk stratification and medication advice.

SUMMARY:
This is an observational clinical study of MRD as a predictor of local treatment in patients with oligometastatic breast cancer. The aim of the study is to assess the correlation between MRD levels and prognosis in patients with oligometastatic breast cancer who have undergone local treatment in order to identify the population that would benefit from local treatment and to develop an individualised treatment plan. Subjects will agree to participate in this study and will be asked to collect as much medical history and demographic information as possible prior to enrolment to confirm that they meet the inclusion/exclusion criteria, and that they will undergo imaging and MRD testing prior to their first study treatment. Furthermore, subjects will undergo tumour imaging and MRD testing every 3 months (±7 days) after MRD treatment for the duration of the study, with additional investigations or more frequent tumour imaging evaluations as clinically indicated during the study.

DETAILED DESCRIPTION:
This is an observational study to investigate the correlation between MRD levels and prognosis in patients with locally treated oligometastases of breast cancer, who have no more than 5 systemic metastases of breast cancer, which may not be confined to the same organ (with the exception of brain metastases), and who have stable systemic control of the disease, and who are to undergo localised treatment. Subjects will read and fully consider the "Informed Consent Form" for this study, sign it in writing if they decide to participate in the study, and complete the Screening Visit no later than 28 days prior to the start of study treatment. For ethical reasons, the screening visit may not be repeated if it was performed prior to the signing of the Informed Consent Form. Subjects were asked to complete imaging and MRD testing prior to their first study treatment, and to undergo on-tumour imaging and MRD testing every 3 months (±7 days) for the duration of the study, and additional investigations or more frequent on-tumour imaging evaluations could be performed during the study based on clinical indications. During this period, subjects continued study treatment until disease progression occurred, toxicity was intolerable, the subject voluntarily withdrew informed consent, or the investigator determined that the subject needed to withdraw from the study. Subjects with disease progression or early withdrawal were also required to complete an exit visit and then enter safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed breast cancer.
2. Previously confirmed metastatic breast cancer by imaging.
3. Eastern Cooperative Oncology Group (ECOG) physical status score of 0-2. (4) Age ≥ 18 years at the time of signing the informed consent form. (5) Subjects willing and able to comply with the study protocol throughout the study period.

(6) Female subjects of childbearing potential must agree to use a highly effective method of contraception during the study.

(7) Voluntarily agree to and sign a written informed consent form and be willing and able to comply with all aspects of the trial protocol, which can be withdrawn by the patient at any time without prejudice.

Exclusion Criteria:

1. Patients with active/refractory infections that require ongoing anti-infective therapy.
2. Severe cardiovascular compromise (history of congestive heart failure greater than New York Heart Association (NYHA) class II), unstable angina or myocardial infarction within the past 6 months, or severe arrhythmia.
3. Subjects with allogeneic organ transplants requiring immunosuppressive therapy. (4) Subjects known to be human immunodeficiency virus (HIV) positive.

5) Subjects with a prior malignancy other than breast cancer, cervical cancer in situ, and non-melanoma skin cancer, unless the prior malignancy has been previously diagnosed and definitively treated for at least 5 years without evidence of subsequent recurrence.

6) Any medical condition that, in the opinion of the Investigator, makes the subject unsuitable for entry into the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The overall study proposes to enrol patients with no more than five lesions of systemic metastases from breast cancer, which may not be confined to the same organ (with the exception of brain metastases), who have stable control of systemic disease, and who are proposed to be treated locally.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
PFS | From enrollment to the end of treatment at 7 months
  It is the time from local treatment of oligometastatic breast cancer to disease recurrence or death from any cause (whichever occurs first)

SECONDARY OUTCOMES:
OS | From enrollment to the end of treatment at 7 months
  It is the period from the date of randomisation until the date of the first confirmation of objective disease progression (as evaluated by the investigator in accordance with RECIST 1.1) or death from any cause (whichever occurs first)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No